CLINICAL TRIAL: NCT06187857
Title: A Feasibility Study of a Virtually Delivered Ecologically Oriented Neurorehabilitation of Memory (EON-MEM) Protocol in Older Adults
Brief Title: A Virtually Delivered Memory Rehabilitation Protocol in Older Adults
Acronym: EONMem_OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham Young University (Other)
Responsible Party: Principal Investigator, Whitney Allen, Principal Investigator, Brigham Young University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EONMem_OA
Record Dates: First submitted 2023-11-27; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Memory Dysfunction; Neurorehabilitation

STUDY DESIGN:
Intervention Model Description: A feasibility study of twenty-five older adults completing the same virtual procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Ecologically Oriented Neurorehabilitation of Memory (EON-Mem) — Feasibility study of a virtually-delivered adaptation of an ecologically oriented neurorehabilitation of memory (EON-Mem) in improving memory for healthy older adults

SUMMARY:
The investigators conducted a feasibility study of a virtually-delivered adaptation of an ecologically oriented neurorehabilitation of memory (EON-Mem) in improving memory for healthy older adults. The primary purposes of this study included determining the feasibility of conducting EON-Mem virtually with older adults and whether a randomized control trial using EON-Mem in older adults is of value.

DETAILED DESCRIPTION:
Twenty-five older adults aged 55 years and older were recruited for participation in the EON-Mem training program adapted and administered virtually. Measures of emotional functioning and cognitive functioning were administered before and following the intervention. Participants attended one virtual treatment session per week for a total of six weeks with daily homework assignments. A priori, feasibility was set at an 80% completion rate. To address questions regarding feasibility, the investigators calculated descriptive statistics on sample information.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 55 and older

Exclusion Criteria:

* Evidence of cognitive dysfunction on the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) as evidenced by a score of 3.3 or more
* History of moderate-to-severe TBI
* History of stroke
* Dementia/neurological diagnoses
* Current chemotherapy or radiation
* Current or history of brain cancer
* Poor sensory function including uncorrected vision, hearing, or speaking impairments that could interfere with learning the intervention, including nonnative English speakers.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Feasibility of study protocols. | Through study completion, an average of 8 weeks.
  To address questions regarding feasibility, the investigators calculated descriptive statistics on sample information and feasibility was set a priori as a completion rate greater than 80% based on previous research.

SECONDARY OUTCOMES:
Memory Outcomes: Repeatable Battery for Neuropsychological Status | Through study completion, an average of 8 weeks.
  To address secondary outcomes, the investigators calculated reliable change indices for memory outcomes on the Repeatable Battery for Neuropsychological Status. The reliable change indices vary from less than -1.96 to greater than 1.96. Greater than 1.96 represents improved memory functioning.
Memory Outcomes: Ecological Memory Simulations | Through study completion, an average of 8 weeks.
  To address secondary outcomes, the investigators calculated reliable change indices for memory outcomes on the Ecological Memory Simulations. The reliable change indices vary from less than -1.96 to greater than 1.96. Greater than 1.96 represents improved memory functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham Young Unversity, Provo, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will be sharing study procedures, study design, and de-identified participant data on the Open Science Framework (OSF).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The dataset will be published in January 2024 and will remain on the website.
URL: https://osf.io/cavkf/?view_only=cc219af15f614756b43742875b6b0b39

REFERENCES:
- Available data/document: Study Protocol — https://osf.io/cavkf/?view_only=cc219af15f614756b43742875b6b0b39

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/57/NCT06187857/Prot_SAP_000.pdf